CLINICAL TRIAL: NCT05035394
Title: A Prospective Randomized Trial Comparing Cataract Surgery as Stand Alone and Cataract Surgery Combined With Kahook Dual Blade Glide Goniotomy or Istent Inject W Trabecular Micro-Bypass Stent in Open-Angle Glaucoma.
Brief Title: Swedish Microinvasive Glaucoma Surgery Study (SMIGS)
Acronym: SMIGS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Anna Barkander, Principal Investigator, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-02970
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Open Angle Glaucoma; Cataract; Kahook Dual Blade Glide; Istent Inject W; MIGS; Goniotomy
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract | interventions — Cataract Extraction; Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cataract surgery as stand alone (Active Comparator): Cataract surgery as stand alone. Cataract surgery will be performed in a standardized fashion.
  Interventions: Procedure: Cataract surgery
- Cataract surgery in combination with Kahook Dual Blade glide goniotomy (Active Comparator): Cataract surgery combined with Kahook Dual Blade Glide goniotomy. The goniotomy will be performed at the end of cataract surgery through the temporal cataract incision.
  Interventions: Procedure: KDB
- Cataract surgery in combination with iStent Inject W implantation (Active Comparator): Cataract surgery combined with iStent Inject W. The two stents will be injected in Schlemms canal at the end of cataract surgery through the temporal cataract incision.
  Interventions: Procedure: Istent

INTERVENTIONS:
Procedure: Cataract surgery — Cataract Surgery in a standardized fashion
  Other Names: Phacoemulsification; Cataract Surgery as stand-alone
  Arms: Cataract surgery as stand alone
Procedure: KDB — Goniotomy with KDB glide will be performed at the end of Cataract Surgery
  Other Names: Kahook Dual Blade Glide, New World Medical, Inc, Rancho Cucamonga, CA; KDB glide
  Arms: Cataract surgery in combination with Kahook Dual Blade glide goniotomy
Procedure: Istent — Two iStent inject W will be injected into Schlemms Canal at the end of Cataract Surgery
  Other Names: iStent inject W; Trabecular Micro-Bypass Stent System Model G2-W, Glaukos Corporation, San Clemente, California
  Arms: Cataract surgery in combination with iStent Inject W implantation

SUMMARY:
The purpose of the study is to investigate the efficacy of Cataract Surgery as stand-alone compared to Cataract Surgery in combination with Kahook Dual Blade Glide goniotomy (KDB) or iStent Inject W Trabecular Microbypass Stent (Istent) in eyes with Open-angle glaucoma.

DETAILED DESCRIPTION:
Glaucoma patients with significant cataract are being informed about the study and potential risks, all participants giving written informed consent and meeting the criteria will become eligibility for study entry. Participants meeting the eligible requirements will be randomized to Cataract Surgery as stand-alone (40 patients) or Cataract Surgery combined with Kahook Dual Blade Glide (40 patients) or iStent Inject W (40 patients).

ELIGIBILITY:
Inclusion Criteria:

* Only one eye per participant
* Clinically significant cataract
* Glaucoma or intraocular hypertension treated with one to four medications and no need for filtering glaucoma surgery at the time of study enrollment.
* Open chamber angle with Schaffer grading three to four in at least two quadrants

Exclusion Criteria:

* Previous glaucoma surgery, including cyclodestructive procedures.
* Selective Laser Trabeculoplasty (SLT) within 90 days prior to planned surgery.
* Exudative age-related macular degeneration, proliferative diabetic retinopathy, clinically significant corneal dystrophy, other eye disease that affect intraocular eye pressure or visual field.
* Unable to participate and make written consent due to another medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in the number of intraocular pressure lowering medications compared to baseline | 12 to 24 months
  Accountability of intraocular pressure lowering medications used by the patient
Number of participants with ≥20 percent intraocular pressure reduction or reduction with ≥1 medication compared to baseline | 12 to 24 months
  Intraocular pressure measured by Goldmann applanation tonometry (GAT)

SECONDARY OUTCOMES:
Number of participants with intraocular pressure ≤21 mm Hg, ≤18 mm Hg, ≤15 mm Hg and ≤12mm Hg | 12 to 24 months
  Intraocular pressure measured by Goldmann applanation tonometry (GAT)

OTHER OUTCOMES:
Number of participants that need further surgery | 12 to 24 months
  Arm comparison of future need for microinvasive surgery, filtering surgery or cyclodestructive laser
Number of participants that need additional medical therapy | 12 to 24 months
  Assessment of the need for future medical therapy in the study groups

CONTACTS AND LOCATIONS:
Overall Officials: Anna Barkander, MD, Principal Investigator — Hospital of Ostersund, department of Ophtalmology
Locations (1):
- Eye clinic at the hospital of Ostersund, Östersund, Östersund, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT05035394/Prot_SAP_000.pdf